CLINICAL TRIAL: NCT02096120
Title: Single Arm Pilot Study of Antimicrobial Treatment of Active Rheumatoid Arthritis Associated With Manifest Periodontitis (Translated From German: Anti-mikrobielle Behandlung Der Aktiven Rheumatoiden Arthritis Bei Manifester Parodontitis - Eine Unkontrollierte Therapie-Pilotstudie)
Brief Title: Full Mouth Disinfection and Antibiotics for Periodontitis in High or Moderate Disease Activity Rheumatoid Arthritis
Acronym: FMD-ABRA
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 130/13; 2439 (Other: Inselspital)
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each 5-10 ml of whole blood, serum and RNA specimen collected in RNA stabilization tubes will be collected at screening and start, and subsequently 1, 3 and 6 months after intervention. Gingival crevicular fluid samples will be collected at start of treatment, after 3 and 6 months.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients

SUMMARY:
The purpose of this study is to determine whether full mouth disinfection in combination with one week antibiotic amoxicillin plus metronidazole antibiotic therapy is improving periodontitis and disease activity of rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a currently incurable disease of unknown origin characterized by joint inflammation and the breakdown of immune tolerance to a variety of antigens, including citrullinated peptides generated by peptidyl-arginine-deiminases (PAD's). Porphyromonas gingivalis (P. g.) derived PAD enzyme (PPAD) citrullinates preferentially C-terminal arginine residues, which may be generated by P.g. derived gingipain protein (Rgpb) cleavage, but several of the originated peptide sequences from enolase, collagen, vimentin or fibrinogen may be cross-reactant to citrullinated RA candidate autoantigens.

Antigen-specific autoantibodies in RA may be present years before clinical disease onset of arthritis, and their precise role in the initiation or perpetuation of the characteristic articular immune processes is currently unclear. The situation for autoantibodies was in similar poorly understood for decades until an unanticipated reduction of RA disease activity could be achieved by therapeutic B cell depletion using anti-CD20 therapy. While anti-CD20 therapy may affect the regeneration of autoantibody producing cells, the investigators aim in the present study to reduce potential oral trigger mechanisms or antigens for cross-reactant autoreactive B cell or plasma cell populations. The study follows the concept of improved RA disease activity by minimization of any inflammatory stimuli associated with periodontitis, e.g. by any underlying microbial colonization, the amount of microbial foreign antigens, achieved by standard oral hygienic means, full mouth disinfection plus adjuvant short term antibiotic therapy in established periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 years or older
* Diagnosis of rheumatoid arthritis according to the ACR/EULAR 2010 classification criteria plus both serological, high titer (>3x ULN) rheumatoid factor and CCP antibody titer
* Severe chronic periodontitis (clinical attachment loss >/= 5mm at two separate locations)
* DAS 28 > 4.2 at screening and inclusion (within 28 days after screening) and 1 out of two additional disease activity criteria:

  1. Synovial hyperplasia >22/66 points on basis of 22 joints, or at least 1/3 of the maximum score when analyzes in at least selected 5 joints of interest OR
  2. Serum CRP > 10 mg/l at screening and at inclusion
* Stable doses for >=3 months, if currently under synthetic or recombinant disease modifying anti-rheumatic drugs. If under anti-CD20 treatment: last rituximab infusion >90 days before inclusion.
* Systemic corticosteroids <= 10 mg and stable for at least 14 days
* Nonsteroidal-antirheumatic drugs and peripheral analgesics at stable doses for at least 14 days

Exclusion Criteria:

* Intolerance to amoxicillin und azithromycin (EBV infection, lymphatic leukemia, exanthema), general hypersensitivity to any beta-lactam antibiotics, intolerance to metronidazole or local anaesthesia
* Current intake of allopurinol or probenicid, oral anticoagulation, disulfiram, phenobarbital phenytoin, lithium or ciclosporin
* Seizures
* Severe cardial electric conduction blockade
* Recent myocardial infraction or instable coronary vessel disease, non-compensated myocardial insufficiency or heart failure
* Non-compensated arterial hypertension
* Genetic cholinesterase deficiency
* General hemorrhagic diathesis or intake of oral anticoagulants
* Intake of monoaminooxidase inhibitors or tricyclic antidepressants
* Liver insufficiency
* Renal failure (eGFR < 30 ml/min)
* Hemoglobin <10 g/dl
* Leukocytes < 3/nl
* Neutrophils < 1/nl
* Platelets < 100/nl
* ALAT oder ASAT > 3x ULN
* Pregnancy or breastfeeding
* Psychiatric or any other condition which could, to the opinion of the investigator, interfere with the compliance of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from inpatient and outpatient hospital rheumatology departments.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-02; Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Improvement in the rheumatoid arthritis disease activity index (DAS28ESR-3v) by >=1.2 points | 3 months
  The DAS28 will be used using 3 variables with 3rd variable erythrocyte sedimentation rate.

SECONDARY OUTCOMES:
Improvement in the rheumatoid arthritis disease activity score (DAS28ESR-3v) by >=1.2 points | At 6 months
Improvement in the rheumatoid arthritis disease activity score when with 3rd variable C reactive protein serum concentration (DAS28CRP-3v) by >=1.2 points | After 3 and 6 months
Improvement in the clinical disease activity index cDAI | After 3 and 6 months
Improvement in the simplified disease activity index cDAI | After 3 and 6 months
Number of patients with 20%, 50% or 70% improvement in the American College of Rheumatology (ACR) response criteria | After 3 and 6 months
Number of patients in ACR/EULAR remission | After 3 and 6 months
% change of B-mode (= gray-scale) and Power-Doppler signals to baseline | After 3 and 6 months
Reduction in the probing pocket depth (PPD) in moderately deep (PPD >/= 4mm) und deep periodontal pockets (PPD > 6mm) | After 3 and 6 months
Improvement in clinical attachment level (CAL), as the sum of PPD plus gingival recession (GR) | After 3 and 6 months
Reduction in the number of sites with bleeding on probing (BoP) | After 3 and 6 months

OTHER OUTCOMES:
Reduction in the number of periodontitis associated microbes on a semi-quantitative level | After 1, 3 and 6 months
  DNA for Porphyromonas gingivalis, Aggregatibacter actinomycetemcomitans, Prevotella intermedia, Fusobacterium nucleatum, Tannerella forsythia, Treponema denticola, Filifactor alocis
Concentration of TNFα, IL-1β, MMP-1 and TIMP-1 1 | After 1, 3 und 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Möller, MD, Principal Investigator — Inselspital, Department for Rheumatology, University of Bern, 3010 Bern, Switzerland
Locations (1):
- Inselspital, Department for Rheumatology, and Dpt. For Periodontology, School for Dentistry, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Aimetti M, Romano F, Guzzi N, Carnevale G. Full-mouth disinfection and systemic antimicrobial therapy in generalized aggressive periodontitis: a randomized, placebo-controlled trial. J Clin Periodontol. 2012 Mar;39(3):284-94. doi: 10.1111/j.1600-051X.2011.01795.x. Epub 2012 Jan 4. PMID 22220822
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Ann Rheum Dis. 2010 Sep;69(9):1580-8. doi: 10.1136/ard.2010.138461. PMID 20699241
- [Background] Klareskog L, Stolt P, Lundberg K, Kallberg H, Bengtsson C, Grunewald J, Ronnelid J, Harris HE, Ulfgren AK, Rantapaa-Dahlqvist S, Eklund A, Padyukov L, Alfredsson L. A new model for an etiology of rheumatoid arthritis: smoking may trigger HLA-DR (shared epitope)-restricted immune reactions to autoantigens modified by citrullination. Arthritis Rheum. 2006 Jan;54(1):38-46. doi: 10.1002/art.21575. PMID 16385494
- [Background] Lundberg K, Kinloch A, Fisher BA, Wegner N, Wait R, Charles P, Mikuls TR, Venables PJ. Antibodies to citrullinated alpha-enolase peptide 1 are specific for rheumatoid arthritis and cross-react with bacterial enolase. Arthritis Rheum. 2008 Oct;58(10):3009-19. doi: 10.1002/art.23936. PMID 18821669
- [Background] de Pablo P, Dietrich T, Chapple IL, Milward M, Chowdhury M, Charles PJ, Buckley CD, Venables PJ. The autoantibody repertoire in periodontitis: a role in the induction of autoimmunity to citrullinated proteins in rheumatoid arthritis? Ann Rheum Dis. 2014 Mar;73(3):580-6. doi: 10.1136/annrheumdis-2012-202701. Epub 2013 Feb 23. PMID 23434568
- [Background] Finckh A, Müller R, Möller B, Dudler J, Kyburz D, Walker UA, et al. Tooth Loss is associated with swollen joints in a cohort of healthy individuals at increased risk of developing RA. European Congress of Rheumatology EULAR 2012. Annals of the rheumatic diseases 2012;71(Suppl).
- [Background] Zandbergen D, Slot DE, Cobb CM, Van der Weijden FA. The clinical effect of scaling and root planing and the concomitant administration of systemic amoxicillin and metronidazole: a systematic review. J Periodontol. 2013 Mar;84(3):332-51. doi: 10.1902/jop.2012.120040. Epub 2012 May 21. PMID 22612369
- [Background] Sampaio E, Rocha M, Figueiredo LC, Faveri M, Duarte PM, Gomes Lira EA, Feres M. Clinical and microbiological effects of azithromycin in the treatment of generalized chronic periodontitis: a randomized placebo-controlled clinical trial. J Clin Periodontol. 2011 Sep;38(9):838-46. doi: 10.1111/j.1600-051X.2011.01766.x. Epub 2011 Jul 19. PMID 21770996
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] Fransen J, van Riel PL. The Disease Activity Score and the EULAR response criteria. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S93-9. PMID 16273792
- [Background] Mandl P, Naredo E, Wakefield RJ, Conaghan PG, D'Agostino MA; OMERACT Ultrasound Task Force. A systematic literature review analysis of ultrasound joint count and scoring systems to assess synovitis in rheumatoid arthritis according to the OMERACT filter. J Rheumatol. 2011 Sep;38(9):2055-62. doi: 10.3899/jrheum.110424. PMID 21885517
- [Background] Aletaha D, Smolen J. The Simplified Disease Activity Index (SDAI) and the Clinical Disease Activity Index (CDAI): a review of their usefulness and validity in rheumatoid arthritis. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S100-8. PMID 16273793
- [Background] Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, Katz LM, Lightfoot R Jr, Paulus H, Strand V, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995 Jun;38(6):727-35. doi: 10.1002/art.1780380602. PMID 7779114
- [Background] Felson DT, Smolen JS, Wells G, Zhang B, van Tuyl LH, Funovits J, Aletaha D, Allaart CF, Bathon J, Bombardieri S, Brooks P, Brown A, Matucci-Cerinic M, Choi H, Combe B, de Wit M, Dougados M, Emery P, Furst D, Gomez-Reino J, Hawker G, Keystone E, Khanna D, Kirwan J, Kvien TK, Landewe R, Listing J, Michaud K, Martin-Mola E, Montie P, Pincus T, Richards P, Siegel JN, Simon LS, Sokka T, Strand V, Tugwell P, Tyndall A, van der Heijde D, Verstappen S, White B, Wolfe F, Zink A, Boers M. American College of Rheumatology/European League against Rheumatism provisional definition of remission in rheumatoid arthritis for clinical trials. Ann Rheum Dis. 2011 Mar;70(3):404-13. doi: 10.1136/ard.2011.149765. PMID 21292833
- [Background] Brulhart L, Zufferey P, Tamborrini G, Möller B, Gerber T, Krebs A, et al. Reproducibility and feasibility of a 22 joints ultrasound score in rheumatoid arthritis: A study among rheumatologists with diverse expertise in musculoskeletal ultrasound. . Annals of the rheumatic diseases 2012;71(Suppl ).
- [Background] Naredo E, Wakefield RJ, Iagnocco A, Terslev L, Filippucci E, Gandjbakhch F, Aegerter P, Aydin S, Backhaus M, Balint PV, Bruyn GA, Collado P, Finzel S, Freeston JE, Gutierrez M, Joshua F, Jousse-Joulin S, Kane D, Keen HI, Moller I, Mandl P, Ohrndorf S, Pineda C, Schmidt WA, Szkudlarek M, Conaghan PG, D'Agostino MA. The OMERACT ultrasound task force--status and perspectives. J Rheumatol. 2011 Sep;38(9):2063-7. doi: 10.3899/jrheum.110425. PMID 21885518
- [Background] Armitage GC. Development of a classification system for periodontal diseases and conditions. Ann Periodontol. 1999 Dec;4(1):1-6. doi: 10.1902/annals.1999.4.1.1. PMID 10863370